CLINICAL TRIAL: NCT04187378
Title: The Effect of Maintenance of Normothermia With Active Warming on Surgical Site Infections in Patients Undergoing Abdominal Surgery
Brief Title: Effect of Active Warming on Surgical Site Infections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Cemile Celebi, M.Sc., Principle Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 31102019-15/III
Record Dates: First submitted 2019-11-26; First posted 2019-12-05 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Surgical Site Infection; Ventral Hernia
Keywords: Hypothermia; Surgical Wound Infection; Herniorrhaphy; Nursing care
MeSH Terms: conditions — Surgical Wound Infection; Hernia, Ventral; Hypothermia

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Control Group (No Intervention): Body temperature of the patients will be measured in the pre-operative service and in the waiting room. Sociodemographic characteristics form, preoperative, intra and postoperative evaluation forms will be completed. Body temperature, blood pressure, respiratory rate, heart rate and O2 saturation of the patients will be monitored every 15 minutes during the operation and postoperative 2 hours and data will be recorded on the data collection form.
- Underbody Blanket Group (Experimental): Patients with hypothermia (<36C) will be warmed by air blown underbody blanket before the surgical procedure. Warming procedure will be continued during and postoperative 2 hours of surgery. Body temperature will be measured by tympanic temperature gauge. Intravenous fluid, antiseptic solutions and irrigation fluids will be given to the patients during surgery by heating before administering. Body temperature, blood pressure, respiratory rate, heart rate and O2 saturation of the patients will be monitored every 15 minutes during the operation and postoperative 2 hours and data will be recorded on the data collection form.
  Interventions: Device: Surgical Underbody Blanket
- Surgical Access Blanket Group (Experimental): Patients with hypothermia (<36C) will be warmed by air blown surgical access blanket before the surgical procedure. Warming procedure will be continued during and postoperative 2 hours of surgery. Body temperature will be measured by tympanic temperature gauge. Intravenous fluid, antiseptic solutions and irrigation fluids will be given to the patients during surgery by heating before administering. Body temperature, blood pressure, respiratory rate, heart rate and O2 saturation of the patients will be monitored every 15 minutes during the operation and postoperative 2 hours and data will be recorded on the data collection form.
  Interventions: Device: Surgical access blanket

INTERVENTIONS:
Device: Surgical Underbody Blanket — Surgical blanket is used to maintain normothermia during abdominal surgery
  Arms: Underbody Blanket Group
Device: Surgical access blanket — Surgical blanket is used to maintain normothermia during abdominal surgery
  Arms: Surgical Access Blanket Group

SUMMARY:
This study evaluates the effect of active warming by maintaining the normothermia during abdominal surgical procedures. The investigators hypothesize that there is no difference in terms of preventing surgical site infections between warm air blown surgical access blanket and underbody blanket.

DETAILED DESCRIPTION:
Hypothermia is defined as a body temperature below 36°C and classified as mild (34°C-36°C), moderate (32°C-33.9°C), severe (<32°C) hypothermia. Hypothermia can be caused by reduced heat production, increased heat loss and / or deterioration of thermoregulation (anesthesia and premedication drugs, antiseptic solutions, low ambient temperature, wet surgical sterile drapes on the patient, use of cold intravenous fluids).

Preoperative, intraoperative and postoperative hypothermia is the drop of body temperature below 36 ° C within one hour before surgery and within 24 hours postoperatively. It is the most common but preventable thermal disorder during anesthesia. It occurs as a result of anesthesia on thermoregulation during surgery and exposure to cold operating room. Although it can be seen in all anesthetized individuals before, during and after surgery due to age, sex, body surface area and body shape; duration, depth, signs and symptoms may vary.

The American Society of Operating Room Nurses (AORN) emphasized the importance of the use of appropriate heating devices in the prevention of hypothermia in surgical patients. Experimental studies and meta-analyzes indicate that active methods of preventing hypothermia (hot air blown systems, hot water circulating blankets and garments, liquid heaters, blood and blood product heaters, etc.), passive methods (wool and synthetic woolen materials, garments and blankets, insulation) materials, etc.) are more effective. It is recommended to use more than one method together to maintain normothermia before, during and after surgery.

Hypothermia is an important problem that should be prevented in surgical patient because it causes serious problems such as delayed wound healing, bleeding, cardiac problems, deterioration of patient comfort, prolonged hospital stay, surgical site infection (SSI) and deaths.

Many guidelines state that the risk of surgical site infection increases three fold due to a decrease in central temperature of 1.9 C. According to the Guidelines for Safe Surgery published by the World Health Organization in 2009; maintaining normothermia during surgery is one of the ten steps intended to reduce the incidence of postoperative surgical site infection. The National Institute for Health and Care Excellence and the Association for Enhanced Recovery After Surgery (ERAS) recommend the maintenance of intraoperative normothermia to prevent surgical site infection.

Surgical nurse; should be aware of the causes of hypothermia and the complications that may occur during the planning, implementation and evaluation of a patient-specific, multi-faceted care; should check the body temperature before, during and after surgery and take precautions to prevent body temperature. Therefore, the body temperature of the patient should be monitored at regular intervals, the body temperature of the preventive interventions must be timely and effective implementation. The maintenance of normothermia in patients with perioperative procedures may reduce the incidence of complications due to hypothermia and may have a positive effect on the success and recovery of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists score I-II-III,
* 18-70 years old,
* Patients undergoing abdominal surgery (ventral hernia)
* Patients whose operation lasts longer than 30 minutes and less than 3 hours

Exclusion Criteria:

* Patients with American Society of Anesthesiologists score IV-V
* Patients with morbid obese (BMI> 40kg / m^2)
* Patients with neurological, psychiatric, neuromuscular disease
* Alcohol and drug addict patients
* Mental retarded patients
* Patients taking medications that affect thermoregulation, such as vasodilators
* Patients with a history of thyroid disease
* Pregnant women
* Patients undergoing pre-intra-post-blood transfusion
* Patients with blood glucose levels above 200 mg / dl

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-08-11 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection Rate | Within the postoperative 30 days
  The rate of surgical site infection will be monitored for each group by the case doctor and principle investigator. The patients will be diagnosed as Surgical Site Infection (SSI) according to CDC Guidelines if there is purulent wound drainage or serous but wound culture is positive within the postoperative 30 days.

SECONDARY OUTCOMES:
Body Temperature | During the surgery and 2 hours after surgery (up to 300 minutes)
  Before surgery, surgical access blanket or underbody blanket will be turned on at the highest temperature of the warming unit ( 43 celsius degree) and the body temperatures will be measured and registered with an tympanic thermometer every 15 minutes during surgery and 2 hours after surgery. Temperatures will be compared with the purposes of determining which one of the two models tested are more effective in keeping patient warm.
Duration of surgery | Day 0 (day of surgery)
  Minutes from skin incision until skin closure

CONTACTS AND LOCATIONS:
Overall Officials: İkbal Çavdar, Professor, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Muğla Sıtkı Koçman University Training and Research Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Batsis JA, Naessens JM, Keegan MT, Huddleston PM, Wagie AE, Huddleston JM. Body mass index and the impact on hospital resource use in patients undergoing total knee arthroplasty. J Arthroplasty. 2010 Dec;25(8):1250-7.e1. doi: 10.1016/j.arth.2009.09.009. Epub 2010 Feb 19. PMID 20171045
- [Background] Bender M, Self B, Schroeder E, Giap B. Comparing new-technology passive warming versus traditional passive warming methods for optimizing perioperative body core temperature. AORN J. 2015 Aug;102(2):183.e1-8. doi: 10.1016/j.aorn.2015.06.005. PMID 26227528
- [Background] Cooper S. The effect of preoperative warming on patients' postoperative temperatures. AORN J. 2006 May;83(5):1073-6, 1079-84; quiz 1085-8. doi: 10.1016/s0001-2092(06)60118-x. PMID 16722285
- [Background] Deren ME, Machan JT, DiGiovanni CW, Ehrlich MG, Gillerman RG. Prewarming operating rooms for prevention of intraoperative hypothermia during total knee and hip arthroplasties. J Arthroplasty. 2011 Dec;26(8):1380-6. doi: 10.1016/j.arth.2010.12.019. Epub 2011 Feb 12. PMID 21316914
- [Background] Hart SR, Bordes B, Hart J, Corsino D, Harmon D. Unintended perioperative hypothermia. Ochsner J. 2011 Fall;11(3):259-70. PMID 21960760
- [Background] Hynson JM, Sessler DI. Intraoperative warming therapies: a comparison of three devices. J Clin Anesth. 1992 May-Jun;4(3):194-9. doi: 10.1016/0952-8180(92)90064-8. PMID 1610573
- [Background] Marino M, Masella R, Bulzomi P, Campesi I, Malorni W, Franconi F. Nutrition and human health from a sex-gender perspective. Mol Aspects Med. 2011 Feb;32(1):1-70. doi: 10.1016/j.mam.2011.02.001. Epub 2011 Feb 26. PMID 21356234
- [Background] Savage JW, Anderson PA. An update on modifiable factors to reduce the risk of surgical site infections. Spine J. 2013 Sep;13(9):1017-29. doi: 10.1016/j.spinee.2013.03.051. Epub 2013 May 24. PMID 23711958
- [Background] Sessler DI. Mild perioperative hypothermia. N Engl J Med. 1997 Jun 12;336(24):1730-7. doi: 10.1056/NEJM199706123362407. No abstract available. PMID 9180091
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- See also: The Essentials of Maintaining Patient Normothermia — https://www.infectioncontroltoday.com/ssi/essentials-maintaining-patient-normothermia
- See also: Peri-operative hypothermia: implications for practice — https://journals.rcni.com/nursing-standard/perioperative-hypothermia-implications-for-practice-ns2013.07.27.45.33.e7742
- See also: Surgical site infections: prevention and treatment — https://www.nice.org.uk/guidance/cg74